CLINICAL TRIAL: NCT02143037
Title: CM Treatment for Alcohol Dependence Using New Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sheila Alessi, Associate Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-040-2; P60AA003510 (NIH)
Record Dates: First submitted 2014-02-24; First posted 2014-05-20 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Alcohol Use Disorder; Contingency Management
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): usual care
  Interventions: Behavioral: usual care
- Experimental Group (Experimental): usual care plus prize contingency management for attending treatment
  Interventions: Behavioral: prize contingency management for attending treatment; Behavioral: usual care

INTERVENTIONS:
Behavioral: prize contingency management for attending treatment
  Arms: Experimental Group
Behavioral: usual care

SUMMARY:
Contingency management (CM) is highly efficacious for reducing substance use, and recent data suggest that reinforcing attendance at treatment can significantly improve treatment outcomes. Importantly, CM interventions that reinforce attendance are more likely to be adopted clinically than those that reinforce abstinence. Having objective indicators of drinking outcomes, nevertheless, is critical for quantifying the benefits of attendance-based CM treatment in alcohol abusing populations. New technology is now available to gauge alcohol use in patients' natural environments. The Secure Continuous Remote Alcohol Monitor (SCRAMx®) continuously monitors alcohol consumption 24 hours a day. As such, it may be ideal for objective evaluation of alcohol consumption during treatment intervention studies, including those that involve CM.

In this study, 114 patients participating in community based outpatient treatment programs for alcohol use disorders will wear SCRAMx for a 12-week period. They will be randomized to standard care or standard care plus CM, with reinforcement contingent upon attendance at treatment. The investigators will assess treatment attendance and alcohol use via SCRAMx and self reports. The investigators expect that patients randomized to the CM intervention will remain in treatment longer and show reductions in both SCRAMx assessed and self reported drinking days relative to those randomized to standard care.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* current diagnosis of alcohol use disorder
* able to pass an informed consent quiz
* agree to wear a SCRAMx monitor for 12 weeks
* have a standard, SCRAMx compatible phone line in their home or agree to attend the clinic at least every other week for data downloads
* agree to sign an off-campus property transfer form and return SCRAMx equipment in 12 weeks

Exclusion Criteria:

* serious, uncontrolled psychiatric illness
* in recovery from pathological gambling
* unstable address
* intend to participate in activities incompatible with SCRAMx in the next 3 months
* are wearing SCRAMx for legal purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
longest duration of actively attending treatment | 3 months
  patient attendance to treatment groups as verified by clinic records (number of days attended out of number of days expected to treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M Alessi, Ph.D., Principal Investigator — UConn Health
Locations (2):
- United States (2):
  - Regional Network of Programs, Inc., Bridgeport, Connecticut
  - Alcohol and Drug Recovery Centers, Inc., Hartford, Connecticut